CLINICAL TRIAL: NCT00722111
Title: Rehabilitation Exercise for Dysphagia Subsequent to Stroke
Brief Title: Exercise for Swallowing Problems After Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: C4796-R
Record Dates: First submitted 2008-07-23; First posted 2008-07-25 (Estimated); Results first posted 2018-03-21 (Actual); Last update posted 2018-03-21 (Actual); Status verified 2018-03

CONDITIONS: Cerebrovascular Accident; Deglutition Disorders
Keywords: tongue; pressure
MeSH Terms: conditions — Stroke; Deglutition Disorders | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Arm 1 (Experimental): lingual press (high-intensity, oral, non-swallowing)
  Interventions: Device: lingual press
- Arm 2 (Experimental): effortful swallowing (high-intensity swallowing)
  Interventions: Behavioral: effortful swallowing
- Arm 3 (Experimental): natural swallowing (high frequency, low intensity swallowing)
  Interventions: Behavioral: natural swallowing
- Arm 4 (Sham Comparator): non-oral sham (control) exercise
  Interventions: Behavioral: non-oral sham (control) exercise

INTERVENTIONS:
Device: lingual press — lingual press (high-intensity, oral, non-swallowing)
  Arms: Arm 1
Behavioral: effortful swallowing — effortful swallowing (high-intensity swallowing)
  Arms: Arm 2
Behavioral: natural swallowing — natural swallowing (high frequency, low intensity swallowing)
  Arms: Arm 3
Behavioral: non-oral sham (control) exercise — non-oral sham (control) exercise
  Arms: Arm 4

SUMMARY:
The purpose of this study is to determine whether stroke patients with swallowing problems will show greater swallowing improvement with intense oral exercise than subjects who perform either a low intensity oral exercise or a sham exercise.

DETAILED DESCRIPTION:
Swallowing problems affect as many as 40% of adults over age 60. Serious consequences are suffered by the numerous patients with neuromuscular deficits secondary to stroke. Patients with dysphagia subsequent to stroke face risk of death from pneumonia, perhaps the most serious sequelae of dysphagia, with malnutrition and dehydration also dire secondary consequences. If stroke patients survive, they require longer hospital stays and nursing home placements with diminished rehabilitation potential. Despite these devastating influences that dysphagia secondary to stroke has on health, evidence supporting the effects of specific interventions on swallowing outcomes in this population is sparse.

Neural plasticity is the mechanism by which the damaged brain relearns "lost behavior" in response to rehabilitation. A goal of this proposal is to implement several principles of exercise and neural plasticity (specificity, repetition, and intensity) in a clinically justifiable manner so they may be used to guide clinical research and ultimately practice. To that end, we will determine how neuromuscular changes affect swallowing outcomes in response to 3 unique 8-week exercise interventions compared with a sham hand (control) exercise group.

The main hypothesis is that after 8 weeks of intense progressive rehabilitation exercise with feedback - lingual press (high-intensity, oral, non-swallowing) stroke patients with dysphagia will show swallowing improvement (defined as an improved score on the Penetration/Aspiration Scale and/or the Residue Scale in the absence of worsening in the other average score) to a greater extent than subjects who perform natural swallowing (low-intensity swallowing) exercises or the sham (control) exercise group. This hypothesis will be tested by 3 discrete objectives: Objective 1: Compare outcomes of four different 8-week exercise interventions among dysphagic stroke patients; Objective 2: Characterize bolus flow, swallowing biomechanics, lingual anatomy and swallowing function of stroke patients through initial calculation of multi-dimensional swallowing profiles pre-intervention and comparison of these profiles post-intervention; and Objective 3: Determine the most appropriate dose of treatment between 4 and 8 weeks for study subjects.

We will randomize 200 men and women post-stroke into four groups (50 subjects per group). Subjects will be randomized into one of four groups, to identify treatment outcomes. The exercise interventions include (a) lingual press (high-intensity, oral, non-swallowing) (b) effortful swallowing (high-intensity swallowing); and (c) natural swallowing (low intensity swallowing), compared with (d) a non-oral sham (control) exercise. All exercises will involve 2 sets of 10 repetitions performed 3 times a day on 3 non-consecutive days per week.

For Objectives 1 and 2 at baseline, week 4, and week 8, each subject will complete simultaneous videofluoroscopic and lingual pressure measures to calculate measures of bolus flow and swallowing biomechanics, which comprise 1) direction (average Penetration/Aspiration Scale Score), completeness (average Residue Scale Score), and duration in msec; 2) isometric and swallowing pressures; and 3) duration and extent of hyolaryngeal excursion and opening of the upper esophageal sphincter. At each of the 3 timepoints, each subject also will complete magnetic resonance imaging (MRI) to measure stroke lesion volume, lingual volume, and lingual tissue differentiation as well as complete swallowing-specific quality of life and dietary questionnaires. For Objective 3, subjects will complete all measures at baseline and weeks 4 and 8 to determine when the most benefits are made during the course of exercise. Knowledge of the dose response will allow for more accurate prescription of the clinical programs.

The Dept. of Veterans Affairs has designated "aging" and its impact on health as high research priorities. As the aging veteran population grows, dysphagia and its deleterious health consequences including pneumonia and/or malnutrition will be an increasing public health burden. In fact, VHA Directive 2006-32 was recently issued (May 17, 2006) defining standard procedures for assessment and treatment of patients with dysphagia. Appropriate diagnosis and treatment for dysphagia with low-cost, non-invasive efficacious exercise programs may not only reduce health care costs, but also will lead to improvements in patient health and quality of life. For patients post-stroke, the implications are enormous when the life-threatening incidence of aspiration is reduced or prevented.

ELIGIBILITY:
Inclusion Criteria:

* 3 months post ischemic or hemorrhagic stroke
* 45 years of age or older
* physician approval of medical stability
* aspiration or penetration of the laryngeal vestibule (score of 3 or higher on Penetration/Aspiration Scale) or post swallow residue in the oropharynx
* able to manage own secretions with no signs of aspiration
* the capacity to provide informed consent

Exclusion Criteria:

* neurologic insult (other than stroke) or neuromuscular disease
* history of radiation to the head or neck
* poorly controlled psychosis
* lack the capacity to complete the exercise program
* refractory alcoholism (on AWD precautions)
* class IV congestive heart failure
* sever chronic obstructive pulmonary disease (home oxygen dependent)
* end-stage renal failure
* allergy to barium (used in radiographic swallowing assessment

Subjects with known contraindication will be excluded from the MRI portion of the protocol:

* Cardiac pacemakers
* Aneurysm clips
* Neurostimulators
* Cochlear implant
* Ossicular prostheses
* Intracranial or intraorbital foreign bodies
* Claustrophobia

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 83 (Actual)
Dates: Start 2011-02; Primary Completion 2011-12 (Actual); Study Completion 2012-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: JoAnne Robbins, PhD, Principal Investigator — Wlliam S. Middleton Memorial Veterans Hospital, Madison
Locations (1):
- Wlliam S. Middleton Memorial Veterans Hospital, Madison, Madison, Wisconsin, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: PI is not available, thus the numbers presented are what was initially entered by research team. From data available, only two of the four treatment arms had subjects randomized to. Thus, for the other treatment arms, no data is available, as PI is not available.
Groups:
- Lingual Strengthening: Isometric Progressive resistance oropharyngeal strengthening for 8 weeks.
- Lingual Pressure Norms: Normative values for lingual pressures
Period: Overall Study
Arm/Group | Lingual Strengthening | Lingual Pressure Norms
Started | 11 | 72
Completed | 11 | 72
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: PI is not available, therefore, no data is available for reporting in this section.Efforts to retrieve data were unsuccessful.
Groups:
- Total: Total of all reporting groups
Arm/Group | Lingual Strengthening | Lingual Pressure Norms | Total
Number analyzed (Participants) | 0 | 0 | 0
Age, Continuous
Sex: Female, Male
Region of Enrollment [unit: participants]

OUTCOME MEASURES:

1. Primary Outcome: Isometric Lingual Pressure
Description: Tongue Strength
Time Frame: 8 weeks
Population: PI is not available, thus the numbers presented are what was initially entered by research team. For the other treatment arms, data is unavailable, as PI is not available. Data was only available for one arm. All efforts were made to retrieve data.
Measure: Mean (Full Range); unit: kPa
Arm/Group | Lingual Strengthening
Number analyzed (Participants) | 11
kPa | 49 [45 to 53]

2. Primary Outcome: Maximum Isometric Tongue Pressure
Description: Peak isometric pressure at 4 sensors
Time Frame: 16 months
Population: PI is not available, thus the numbers presented are what was initially entered by research team. For the other treatment arms, data is unavailable, as PI is not available.Data was only available for two arms. All efforts were made to retrieve data.
Measure: Mean (Full Range); unit: kPa
Arm/Group | Lingual Strengthening | Lingual Pressure Norms
Number analyzed (Participants) | 11 | 72
kPa | 49 [45 to 53] | 78 [5 to 270]

ADVERSE EVENTS:
Description: PI is not available, thus it is impossible to determine if Adverse Events were collected or assessed. All efforts were made to retrieve data.
Arm/Group | Lingual Strengthening | Lingual Pressure Norms
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes